CLINICAL TRIAL: NCT01190657
Title: A Multiple-center, Self-controlled Open Study to Evaluate Efficacy and Safety of Teprenone in Patients With Acute Gastritis, Acute Gastric Lesion of Chronic Gastritis With Acute Exacerbation or Gastric Ulcer
Brief Title: Efficacy and Safety of Teprenone in Patients With Acute Gastritis, Acute Gastric Lesion of Chronic Gastritis With Acute Exacerbation or Gastric Ulcer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P216
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Last update posted 2013-04-01 (Estimated); Status verified 2013-03

CONDITIONS: Acute Gastritis; Gastric Ulcer
Keywords: Teprenone; safety; efficacy; acute gastric lesion; chronic gastritis
MeSH Terms: conditions — Stomach Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Selbex 50mg (14 days) (Experimental)
  Interventions: Drug: Selbex
- Selbex 50mg (56 days) (Experimental)
  Interventions: Drug: Selbex

INTERVENTIONS:
Drug: Selbex — 50mg/day, 3 times/day, for 14 days
  Arms: Selbex 50mg (14 days)
Drug: Selbex — 50mg/day, 3 times/day, for 56 days
  Arms: Selbex 50mg (56 days)

SUMMARY:
This is a self-controlled, open, multiple-center clinical trial.

ELIGIBILITY:
Inclusion criteria

1. Age is over 18 years old , men or women
2. Erosive lesions or flat lesions with thin white coating in acute gastritis, acute stage of chronic gastritis with over three lesions (including three lesions) by endoscopy prior to study in 3 days or diagnosed by clinical symptoms and signs;
3. Signed the informed consent forms.

Exclusion criteria

1. Patients without inclusion criteria
2. Patients with significant cardiovascular, pulmonary, hepatic, renal or hemopoietic system primary disease
3. Patients with other digestive diseases.
4. Patients with operation on stomach and duodenum.
5. Patients administered with nonsteroidal anti-inflammatory drugs (NSAIDs) and corticosteroids
6. Patients with severity trauma, surgery, infection and shock.
7. Patients with any kind of tumor
8. Women either pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1184 (Actual)
Dates: Start 2010-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Endoscopic results of ulcer lesion | 56 days
  Heal rate = (healed cases + significant improved cases)/total cases administered ×100 %
Total effective rate | 56 days.
  Total effective rate = (healed cases + significant improved cases + effective cases)/total cases administered ×100 %.

SECONDARY OUTCOMES:
Symptoms improved level | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Yaozong Yuan, Principal Investigator — Ruijin Hospital
Locations (26):
- China (26):
  - Chinese People's Liberation Army General Hospital of Beijing Military, Beijing
  - Chongqing First People's Hospital, Chongqing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Wuhan Union Hospital, Hubei
  - Changsha Central Hospital, Hunan
  - Hunan Provincial People's Hospital, Hunan
  - Nanjing First Hospital, Jiangsu
  - Nanjing General Hospital of Nanjing Military Command, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Jiangsu
  - The Second Affiliated Hospital of Suzhou University, Jiangsu
  - Wuxi #2 People's Hospital, Jiangsu
  - Jilin University First Hospital, Jilin
  - Shengjing Hospital of China Medical University, Liaoning
  - Shanghai Changzheng Hospital, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - Shanghai Renji Hospital, Shanghai
  - Shanghai Ruijin Hospital, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai
  - Shanxi Provincial People's Hospital, Shanxi
  - The Second Affiliated Hospital of the Medical College of Xi'an Jiaotong University, Shanxi
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Sichuan
  - The Affiliated Hospital of Luzhou Medical College, Sichuan
  - Tongji Hospital, Sichuan
  - Hangzhou Red Cross Hospital, Zhejiang
  - The First Affiliated Hospital of Zhejiang University, Zhejiang